CLINICAL TRIAL: NCT05834361
Title: The Administration Time Point of Carboprost Methylate and Effects on Perioperative Complications and Cervical Ripening Effect in Artificial Abortion
Brief Title: The Time Point of Carboprost Methylate Administration and Perioperative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K23C0074
Record Dates: First submitted 2023-04-05; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-01

CONDITIONS: Artificial Abortion, PONV(Post Operative Nausea and Vomiting)
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- early administration of carboprost methylate (Experimental): Shortening the vaginal administration time of carboprost methylate, approximately 20 minutes before the surgery. Carboprost methylate was given when patients enter the operation room area.
  Interventions: Drug: early vaginal administration of carboprost methylate
- delayed administration of carboprost methylate (Active Comparator): Delay the vaginal administration time of carboprost methylate, approximately 2 hours before the surgery. Carboprost methylate was given when patients were in the ward.
  Interventions: Drug: delayed vaginal administration of carboprost methylate

INTERVENTIONS:
Drug: early vaginal administration of carboprost methylate — In this group, the administration time point of carboprost methylate is 20 minutes before the surgery.
  Arms: early administration of carboprost methylate
Drug: delayed vaginal administration of carboprost methylate — In this group, the administration time point of carboprost methylate is usually 110-120 minutes before the surgery.
  Arms: delayed administration of carboprost methylate

SUMMARY:
Artificial abortion is the most widely used procedure in termination of first-trimester pregnancy. Cervical ripening before the operation guarantees operative convenience and decreases complications. An overstrained cervical dilation associates with uterine perforation, cervical laceration and cervical incompetence. To address the issue, various mechanical and pharmaceutical methods have been applied to prepare the cervix before transvaginal procedures. Prostaglandin analogues (PGs) play an important role in ripening the cervix or promoting uterine contraction in gynecology and obstetrics. As most tissues express prostaglandin receptors, vomiting, nausea, fever, diarrhea and abdominal pain can hardly be avoided with PGs administration. Longer PGs action contributes to better cervical ripening, but more uncomfortableness at the same time. These annoying symptoms may affect the participants' satisfaction and increase perioperative risks. To balance the safety and effectiveness of the surgery as well as patients' feeling, a proper timing for cervical ripening should be investigated. However, the administration timing of PGs has not reached a broad consensus, ranging from 16 hours to 2 hours before surgery. Carboprost methylate (CM), a PG-F2α analogue, has been used nationwide for cervical ripening in China. To minimize the side effects of PGs without affecting cervical ripening, the investigators intended to explore shortening the action time of CM in cervical preparation before artificial abortion. Thus, the investigators conducted this prospective cohort study and aimed to examine the efficacy of early and delayed vaginal administration of CM before surgery, and optimized both the perioperative safety and participants' convenience. The investigators hypothesize that early vaginal administration of CM would not affect the cervical ripening status, but will greatly reduce the unpleasant complications among the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-59
* Signed informed consent.
* Admitted to hospital for surgical termination of unplanned pregnancy
* Gestational weeks range between 7 to 10
* Average diameter of the gestational sac was no larger than 4cm

Exclusion Criteria:

* Massive vaginal bleeding
* Severe abdominal pain at admission (numerical rating scale, NRS>3)
* Genital tract infection
* Contraindication of PGs (including uncontrolled hypertension, asthma, glaucoma, severe heart disease or allergy to prostaglandins, etc.)
* Prior history of vaginal delivery

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Total adverse events | Baseline (Before surgery)
  total adverse events before anesthesia, including abdominal pain, nausea, vomiting, defecate desire and diarrhea.

SECONDARY OUTCOMES:
Numerical rating scale (NRS) before surgery | Baseline (Before surgery)
  NRS score before surgery (score from 0-10)(0 = no pain; 10 = worst pain imaginable)
Postoperative nausea and vomiting (PONV) | 4 hours after surgery
  The pond percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen RH, Goldberg AB. Cervical dilation before first-trimester surgical abortion (<14 weeks' gestation). Contraception. 2016 Apr;93(4):277-291. doi: 10.1016/j.contraception.2015.12.001. Epub 2015 Dec 9. PMID 26683499
- [Background] Pierce S, Bakker R, Myers DA, Edwards RK. Clinical Insights for Cervical Ripening and Labor Induction Using Prostaglandins. AJP Rep. 2018 Oct;8(4):e307-e314. doi: 10.1055/s-0038-1675351. Epub 2018 Oct 29. PMID 30377555
- [Background] Hwang JY, Song SH. Optimal Dose of Vaginal Misoprostol for Cervical Ripening before Hysteroscopy: A Randomized Double-Blind Study. J Minim Invasive Gynecol. 2018 Sep-Oct;25(6):1031-1034. doi: 10.1016/j.jmig.2018.01.022. Epub 2018 Jan 31. PMID 29409965
- [Derived] Zhao Y, Xue W, Chen W, Zhang D. Delayed Administration of Carboprost Methylate Reduces Perioperative Complications Without Affecting Cervical Ripening Effect in Surgical Abortion: A Randomized Controlled Trial. J Obstet Gynaecol Res. 2025 Oct;51(10):e70107. doi: 10.1111/jog.70107. PMID 41088336